CLINICAL TRIAL: NCT03998397
Title: Self-estimates and Objective Measurement of Blood Alcohol Concentration in Patients With Alcohol Intoxication Presenting to an Emergency Department
Brief Title: Self-estimates and Objective Blood Alcohol Concentration in Emergency Department
Acronym: SEOBACED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2018_843_0009
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder; Blood Alcohol Content
Keywords: blood alcohol concentration; Emergency Department; Alcohol use disorders
MeSH Terms: conditions — Alcoholism; Emergencies | interventions — Blood Specimen Collection; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with alcohol use disorders (Experimental)
  Interventions: Biological: blood alcohol concentration withdrawal
- patients without alcohol use disorders (Experimental)
  Interventions: Biological: blood alcohol concentration withdrawal

INTERVENTIONS:
Biological: blood alcohol concentration withdrawal — The blood alcohol concentration is systematically performed in all intoxicated patients admitted in Emergency Department

SUMMARY:
Many patients presenting in Emergency Department (ED) present alcohol acute intoxication. Some previous studies in general population found that young people under- or over-estimated of blood alcohol concentration (BAC). The hypothesis of the study is that self-estimation of BAC by the patient is under-estimated. Moreover, comparing self-estimation of BAC and objective measure of BAC, which is routinely performed in ED, could increase in patients the awareness of the disorders, increase motivation to change of the patient, and increase the rates of seeking-treatment six months after the first evaluation, in particular in patients with alcohol use disorders.

To the investigators knowledge, there is no study investigating self-estimation, compared to objective measurement of blood alcohol concentration in patients with alcohol intoxication presenting to an Emergency Department (ED). The study will assess blood alcohol concentration and self-estimates of BAC, using the Subjective Effects of Alcohol Scale for Measuring Subjective Response to Alcohol in 100 patients with or without alcohol use disorders according to DSM-5 classification (using MINI scale and Alcohol Use Disorders Identification Test (AUDIT)

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in Emergency Department while intoxicated will be included in the study, including patients with or without alcohol use disorders according to DSM-5 classification.
* aged 15-64 years old
* patients who will be orally informed and receive a written summary
* blood alcohol concentration of 60mg/dl or higher
* Patients not opposed to participating in the study, who have received an oral and written information

Exclusion Criteria:

* Drug intoxication (cannabis, opiates, amphetamines, cocaine), psychotropic medication intoxication (benzodiazepines, antipsychotics), primary neurologic conditions, mental retardation, dementia, amnestic disorders, mental disorders due to a general, medical condition and substance-induced psychotic disorders.

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Mean change between real blood alcohol concentration and self-estimated blood alcohol concentration | Day =0 (day of patient inclusion)
  Comparison of real blood alcohol concentration and self-estimated blood alcohol concentration

SECONDARY OUTCOMES:
Mean change between real blood alcohol concentration and self-estimated blood alcohol concentration in patient with alcohol use disorders | Day =0 (day of patient inclusion)
  Comparison of real blood alcohol concentration and self-estimated blood alcohol concentration with alcohol use disorders according DSM-5 classification (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
Mean change between real blood alcohol concentration and self-estimated blood alcohol concentration in patient without alcohol use disorders | Day =0 (day of patient inclusion)
  Comparison of real blood alcohol concentration and self-estimated blood alcohol concentration without alcohol use disorders according DSM-5 classification (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
Measure motivation to change during the first interview at the Emergency Department | Day =0 (day of patient inclusion)
  Measure motivation to change during the first interview at the Emergency Department
Measure motivation to change six months following the first interview at the Emergency Department | six months following the first interview at the Emergency Department
  Measure motivation to change six months following the first interview at the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Alain Dervaux, Pr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DOI:10.1016/j.euroneuro.2020.09.032 November 2020European Neuropsychopharmacology 40(4):S20 P.029 Self-estimation of blood alcohol concentration in patients admitted for acute alcohol intoxication in emergency department